CLINICAL TRIAL: NCT03125135
Title: Accuracy of Noninvasive Pulse Oximeter Sensor (MightySat RX)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TR27761-TP16850A
Record Dates: First submitted 2017-04-14; First posted 2017-04-24 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Test Subject (Experimental): All subjects are enrolled into the test group and all subjects receive the MightySat RX Pulse Oximeter Sensor.
  Interventions: Device: MightySat RX Pulse Oximeter Sensor

INTERVENTIONS:
Device: MightySat RX Pulse Oximeter Sensor — Noninvasive pulse oximeter finger sensor.

SUMMARY:
In this study, the level of oxygen within the blood will be reduced in a controlled manner by reducing the concentration of oxygen the study volunteer breathes. The accuracy of a noninvasive pulse oximeter sensor will be assessed by comparison to the oxygen saturation measurements from a laboratory blood gas analyzer.

ELIGIBILITY:
Competent non-smoking adults

Inclusion Criteria:

* Subjects must understand and consent to be in the study.
* American Society of Anesthesiology Class 1 (Healthy subjects without any systemic disease at all).

Exclusion Criteria:

* Subjects who have any systemic disease at all.
* Subjects who do not understand the study and the risks.
* Smokers.
* Subjects who are pregnant.
* Subjects having either signs or history of peripheral ischemia.
* Others deemed ineligible by the clinical staff.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2014-11-12 (Actual); Primary Completion 2014-12-17 (Actual); Study Completion 2014-12-17 (Actual)

PRIMARY OUTCOMES:
Accuracy of Sensor | 1-5 hours
  Accuracy will be determined by comparing the noninvasive blood oxygen saturation measurement of the pulse oximeter to that obtained from a blood sample and calculating the arithmetic root mean square error (Arms) value.
Accuracy of Sensor during motion | 1-5 hours
  Accuracy will be determined by comparing the noninvasive blood oxygen saturation measurement of the pulse oximeter to that obtained from a blood sample during motion conditions and calculating the arithmetic root mean square error (Arms) value.

CONTACTS AND LOCATIONS:
Locations (1):
- Masimo Corporation, Irvine, California, United States